#### **CLINICAL STUDY PROTOCOL**

A Randomized, Double-Masked, Parallel Group, Multicenter, Study to Evaluate Efficacy and Safety of SPARC's SDN-037 Twice Daily Compared with Vehicle for The Treatment of Inflammation and Pain Associated with Ocular Surgery.

Protocol No. : CLR\_16\_31

**Protocol Version**: Version 01 Amendment 03

Protocol Date : 22JAN2020

Plan Version No. : 1

Plan Version Date : 17SEP2020

### **SIGNATURE PAGE**





#### STATISTICAL ANALYSIS PLAN DETAILS

| TRIAL FULL TITLE | A Randomized, Double-Masked, Parallel Group, Multicenter,<br>Study to Evaluate Efficacy and Safety of SPARC's SDN-037 |
|---|---|
| | Twice Daily Compared with Vehicle for The Treatment of |
| | Inflammation and Pain Associated with Ocular Surgery |
| CT IDENTIFIER | NCT03426267 |
| SAP VERSION | 1 |
| SAP VERSION DATE | 17SEP2020 |
| TRIAL CHIEF | MULTI-CENTER |
| INVESTIGATOR | |





#### 2 ABBREVIATIONS AND DEFINITIONS

| ACC | Anterior Chamber Cell |
|--------|----------------------------------------------|
| ACF | Anterior Chamber Cen |
| AE | Adverse Event |
| BCVA | Best Corrected Visual Acuity |
| BID | Twice a day (bis in die) |
| BSCVA | Best-Spectacle Corrected Visual Acuity |
| CI | Confidence Interval |
| CRO | Contract Research Organization |
| eCRF | electronic Case Report Form |
| ETDRS | Early Treatment Diabetic Retinopathy Study |
| FDA | Food and Drug Administration |
| GCP | Good Clinical Practice |
| GLP | Good Laboratory Practice |
| IB | Investigator's Brochure |
| ICF | Informed Consent Form |
| ICH | International Council for Harmonisation of |
| | Technical Requirements for Pharmaceuticals |
| | for Human Use |
| IEC | Independent Ethics Committee |
| IND | Investigational New Drug |
| IOP | Intraocular Pressure |
| IOL | Intra Ocular Lens |
| IP | Investigational Product |
| IRB | Institutional Review Board |
| IWRS | Interactive Web Response System |
| mITT | Modified Intent-To-Treat |
| LAR | Legally Acceptable Representative |
| LOCF | Last Observation Carried Forward |
| logMAR | Logarithm of the Minimum Angle of |
| | Resolution |
| MedDRA | Medical Dictionary for Regulatory Activities |
| NDA | New Drug Application |
| OPD | (in-)Office Physician Dispensing |
| PP | Per Protocol |
| PT | Preferred Term |
| RLD | Reference Listed Drug |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |

| SPARC | Sun Pharma Advanced Research Company, |
|--------|-------------------------------------------|
| | Ltd. |
| SUSAR | Suspected Unexpected Serious Adverse |
| | Reaction |
| TEAE | Treatment-Emergent Adverse Event |
| VAS | Visual Analog Scale |
| WHO-DD | World Health Organization Drug Dictionary |
| w/v | Weight/Volume |

### 3 SUMMARY OF LIST OF CHANGES FROM PROTOCOL





#### 4 INTRODUCTION

| 4.1 Preface |
|---|
| Sun Pharma Advanced Research Company Ltd. (SPARC) has developed a novel topical ophthalmic |
| formulation of difluprednate as a for the treatment of |
| inflammation and pain associated with ocular surgery. SPARC intends to develop the ophthalmic difluprednate product at a dose dose and with a dose |
| difluprednate product at a dose and with a dose and with a dose and with a dose |
| 4.2 Purpose of the analyses |
| These analyses will assess the efficacy and safety of topical administration of |
| 5 STUDY OBJECTIVES AND ENDPOINTS |
| 5.1 Study Objectives |
| To evaluate the efficacy and safety of topical administration of |
| dose after surgery followed by |
| 5.2 Endpoints |
| Efficacy: |
| The primary efficacy endpoint is the proportion of subjects with an ACC grade of 0 at Day 15 |
| The key secondary efficacy endpoint is the proportion of subjects who achieve a pain score of 0 at Day 15 |
| at Day 15. |
| • |

#### 6 STUDY METHODS

#### 6.1 General Study Design and Plan

 This study is a phase 3, randomized, multicenter, double-masked, vehicle-controlled, parallelgroup clinical study.

| • | Type of control: |
|---|---|
| • | Level and method of blinding: |
| • | <b>Method of treatment assignment</b> : Subjects who qualify via inclusion and exclusion criter will be assigned to study treatment groups assigned. |
| • | assigned to study treatment groups. |
| • | |
| • | |
| | · |
| 2 Inc | clusion-Exclusion Criteria and General Study Population |
| • | INCLUSION CRITERIA 1. Be male or female, of 18 years of age or older |
| | 5. Able to self-instill the IP or have a caregiver available to instill all doses of the IP, as instructed |

6. Females of childbearing potential must not be pregnant (as confirmed by a negative urine pregnancy test

7. Be able and willing to follow study instructions and complete all required visits

#### • EXCLUSION CRITERIA

1. Any known allergy or hypersensitivity to difluprednate therapy





#### **6.4 Study Termination**

The study may be stopped at any time by the sponsor, the investigator and/or the IRB with appropriate notification.

If the study is prematurely terminated or suspended for any reason, the investigator/institution should promptly inform the subjects, should assure appropriate therapy and follow-up for the subjects, and, where required by the applicable regulatory requirement(s), should inform the regulatory authority(ies).

















Page **19** of **34** 









| <u> </u> |
|---|
| 10 EFFICACY ANALYSIS |
| 10.1 Primary Efficacy Analysis |
| The primary efficacy endpoint is the proportion of subjects with an ACC grade of 0 at Day 15 |
| The primary emeacy enapoint is the proportion of subjects with an Ace grade of 6 at buy 15 |





| 11.5 Relationship of Treatment-Emergent Adverse Events to the IP A summary of TEAEs by SOC, PT, and relationship to the IP will be presented by treatment group. The relationships indicate the investigator's assessment of whether or not the event was caused by the IP. The possible relationships are "Unrelated", "Unlikely", "Possibly", "Probably", and "Certainly". |
|---|
| <b>11.6 Serious Adverse Events</b> Serious adverse events (SAEs) will be listed by subject; SAEs will be summarized by event and treatment group. |
| 11.7 Adverse Events Leading to Study Drug Withdrawal All AEs leading to study withdrawal or study drug withdrawal will be listed and summarized. |



#### 12 REPORTING CONVENTIONS

Summary tables and listings (e.g., post text tables and individual subject data listings are prepared according to ICH Guideline E3) include a header, showing Protocol Number, Status, and sponsor; and a "footer" providing explanatory notes that indicate as a minimum:

- SAS program name and data file source
- Date of data extraction
- Date of output generation

Post text tables also include reference(s) to the subject data listing(s) that supports the summary data. The data extraction date links the output to the archived database that is locked to ensure the replication of the results.

Post text tables will be organized with respect to treatment groups for safety and efficacy. The order of presentation will be chronological for visits. A total column will appear as the last column, as applicable. The summary tables clearly indicate the number of subjects to which the data apply and unknown or not performed are distinguished from missing data.

Summary tables for medications and medical conditions are coded according the WHO Drug Dictionary and MedDRA respectively. Adverse event preferred terms and body/organ systems are coded using the MedDRA dictionary. The MedDRA dictionary can be used, as well, in the coding of signs and symptoms, medical history, physical examination abnormalities, and clinical diagnoses.

Supportive individual subject data listings, at a minimum, are sorted and presented by subject ID and treatment. Listings also include visit number, visit date, and days relative to the initiation of treatment.



















| · |
|---|